CLINICAL TRIAL: NCT06551857
Title: The Effect of Cancer Treatments on Speech Perception in Noise, Cognition, and Hearing-Related Quality of Life
Acronym: CaSPiN
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tytti Willberg, Principal Investigator, Turku University Hospital
Other Study IDs: T1700/2024; 2024-513437-21-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-03; First posted 2024-08-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Hearing Loss Ototoxic; Cognitive Decline; Quality of Life
Keywords: speech perception in noise; ototoxicity; hearing loss; cancer; cisplatin; oxaliplatin; cognition
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Ototoxicity; Hearing Loss | interventions — Drug Therapy; Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cisplatin: 50 patients receiving cisplatin as the standard care for their underlying malignancy
  Interventions: Other: Chemotherapy, chemoradiation, radiation therapy
- Cisplatin-based chemoradion therapy in the head and neck region: 50 patients receiving cisplatin-based chemoradiation therapy in the head and neck region as the standard care for their underlying malignancy
  Interventions: Other: Chemotherapy, chemoradiation, radiation therapy
- Head and neck region radiation therapy: 50 patient receiving head and neck region radiation therapy as the standard care for their underlying malignancy
  Interventions: Other: Chemotherapy, chemoradiation, radiation therapy
- Oxaliplatin: 50 patients receiving oxaliplatin as the standard care for their underlying malignancy
  Interventions: Other: Chemotherapy, chemoradiation, radiation therapy
- Control: 50 healthy volunteers who have never received any ototoxic medications

INTERVENTIONS:
Other: Chemotherapy, chemoradiation, radiation therapy — Cancer treatment
  Groups: Cisplatin; Cisplatin-based chemoradion therapy in the head and neck region; Head and neck region radiation therapy; Oxaliplatin

SUMMARY:
The study will assess the effect of cancer treatments on speech perception in noise, cognition, and hearing-related quality of life by monitoring 200 cancer patients receiving standard care for their underlying malignancy.

DETAILED DESCRIPTION:
The study will assess the effects of four different types of cancer treatments on speech perception in noise, hearing thresholds, cognition, and hearing-related quality of life over a follow-up period of 3 years.

The speech perception in noise will be assessed using the Finnish matrix sentence test. Other hearing measures include transient and distortion product otoacoustic emissions, impedance audiometry and pure-tone audiometry extending to high frequencies (0.125kHz - 16kHz).

Hearing-related quality of life will be assessed using Speech, Spatial, and Qualities 12 -questionnaire, Vanderbilt Fatigue Scale 10 -questionnaire and Tinnitus Handicap Index. Cognitive functions will be assed using Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire and neuropsychological tests. The neuropsychological tests included in the study are Continuous Performance Test, Continuous Auditory Test of Attention, Trail Making Test A & B, Stroop Test, Coding and Digit span tasks from the Wechsler Adult Intelligence Scale - Fourth Edition, Word List task from Wechsler Memory Scale III, and Controlled Oral Word Association Test.

Neuropsychological assessments will be conducted at baseline and 1 year and 3 years after the end of the treatments. All other assessments will be conducted at baseline and at 3-4 months, 1 year, and 3 years after the end of the initial treatments.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* native Finnish speaker
* age-normative hearing
* for participants in the treatment arms: diagnosis of a malignancy that will be treated with curative intent with any of the following: 1) Cisplatin as the main chemotherapeutic agent, 2) oxaliplatin as the main chemotherapeutic agent, 3) cisplatin-based chemoradiation therapy in the head and neck region, 4) radiation therapy in the head and neck region

Exclusion Criteria:

* inability to provide written informed consent
* Current or prior major otological condition that has affected or has had the potential to affect hearing
* Conductive or asymmetric sensorineural HL of any severity
* Severe sensorineural HL
* Prior malignancy treated with chemotherapeutics or radiation therapy
* Prior use of ototoxic medications
* Any significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk by participation in the trial, or may influence the result of the trial.
* Any condition that, in the opinion of the investigator, would interfere with adherence to the trial requirements.

For participants in the treatment arms:

* Allergy or hypersensitivity to trial medications or their ingredients
* Pregnancy or breast-feeding, aim of becoming pregnant during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 patients diagnosed with a malignancy that will be treated with curative intent using one of the treatment modalities under investigation (50 patients / group). The study will also include a control group of 50 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Speech perception in noise | 4 months
  The treatment-related change in speech perception in noise (in decibel signal-to-noise ratio (db SNR)) from baseline to first follow-up at 3-4 months after the end of the treatment.

SECONDARY OUTCOMES:
Long-term effects on speech perception in noise | 3 years
  Treatment-related long-term changes in speech perception in noise (in decibel signal-to-noise ratio (dB SNR)) measured with the Finnish matrix sentence test
Short- and long-term effects on high frequency hearing | 3 years
  Treatment-related changes in high frequency (8-16kHz) hearing thresholds
Hearing-related quality of life - Sound quality | 3 years
  Treatment-related changes in hearing related quality of life measured using the total score from Speech, Spatial, and Qualities 12 question questionnaire (SSQ-12). Responses are given with a VAS scale from 0 to 10, with 10 indicating perfect hearing performance and 0 worst possible performance. Range for total scores is 0-120, and decrease in scores indicates deterioration in hearing-related quality of life.
Hearing-related quality of life - Fatigue | 3 years
  Treatment-related changes in hearing-related fatigue are measured using the total score from Vanderbilt Fatigue Scale for Adults (10 question version, VFS-A-10). Responses are given in a 5-point Likert scale. The range for total scores is 0-40 with higher scores indicating more fatigue / worse score. An increase in the total score indicates increased listening-related fatigue.
Hearing-related quality of life - Tinnitus | 3 years
  Treatment-related changes in tinnitus symptoms are measured using the total score from Tinnitus Handicap Inventory (THI). The questionnaire provides a total score between 0 and 100, with larger score indicating more tinnitus-related handicap. An increase in the total score indicates increased tinnitus-related handicap.
Treatment-related changes in brain glucose metabolism | 3 years
  Treatment-related brain changes are evaluated from the FDG PET by assessing the voxel-wise mean change in the standardized uptake value ratios (SUVRs) from baseline to follow-up. Decrease in SUVRs indicates treatment-related decrease in brain glucose metabolism.

OTHER OUTCOMES:
Treatment-related changes in cognition | 3 years
  Treatment-related changes in cognition are evaluated using the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) questionnaire. Responses are given in a five-point Likert-type scale and are presented as subscale scores for four domains: perceived cognitive impairments, impact of perceived cognitive impairments on quality of life, comments from others, and perceived cognitive abilities. Higher score indicates better perceived performance.

CONTACTS AND LOCATIONS:
Overall Officials: Tytti Willberg, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No
The data is collected from a clearly specified patient population and includes personal information that can be used to identify individual participants, even after pseudonymization. Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and Analytic Code will be shared through Open Science Framework immediately following publication and be available with no end date.